CLINICAL TRIAL: NCT05999162
Title: Changing Patterns and Surgical Outcomes for Mechanical Ileus in the Era of Minimally Invasive Colorectal Surgery
Brief Title: Mechanical Ileus in the Era of Minimally Invasive Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202306117RINA
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer; Adhesion
Keywords: adhesive ileus; internal herniation; colorectal cancer; minimally invasive surgery
MeSH Terms: conditions — Colorectal Neoplasms; Tissue Adhesions | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally invasive surgery (MIS): The patients underwent minimally invasive surgery for the treatment of colorectal cancer.
  Interventions: Procedure: Minimally invasive surgery
- Traditional open surgery (TOS): The patients underwent traditional open surgery for the treatment of colorectal cancer.

INTERVENTIONS:
Procedure: Minimally invasive surgery — Minimally invasive surgery includes laparoscopic surgery or robotic surgery for the treatment of colorectal surgery.
  Groups: Minimally invasive surgery (MIS)

SUMMARY:
The present study was to investigate if the incidence, patterns and surgical outcomes of mechanical ileus have changed in the era of minimally invasive surgery (MIS).

DETAILED DESCRIPTION:
Mechanical ileus, generally caused by post-operative bowel adhesion, represented 12-16% of emergency surgical admissions and 20% of emergency surgical procedures. Opening the peritoneal cavity, in whatever type of surgery, leads to the formation of potentially obstructive structures (adhesions or bands) in almost 95% of patients. The adhesion resulted from the irritation of the peritoneum caused by surgical trauma or intra-abdominal infection. Bowel adhesions can lead to clinical manifestations within a few weeks or even several years after the surgery. It has been reported that traditional open surgery (TOS) for colorectal cancer were associated with a particularly higher risk of adhesion formation and related complications. Within two years after colorectal surgery, 14.3% of the patients will suffer from small bowel obstruction, and 2.6% will require a surgical intervention for the treatment of this obstruction, and this incidence is even higher after rectal surgery. Adhesive ileus has been a clinical conundrum. Overall, nearly one-fifth of patients needed re-admission for a recurrent disease, even they had been successfully treated by surgical, or non-surgical methods during the index admission.

During the last decade, minimally invasive surgery (MIS), either via laparoscopic or robotic approach, has become the standard procedures for the treatment of colorectal cancer. Theoretically, MIS is associated with a much lower rate of postoperative formation of adhesions than TOB, since adhesion formation represents a stepwise failure of peritoneal tissue repair mechanisms, which can be prevented by the clean dissection, minimal blood loss and/or less-environmental exposure of the bowel inherent in MIS. Some researchers supported this concept by showing MIS colorectal surgery is associated with fewer adhesion-related admissions than open surgery. However, most reported case series were retrospective uncontrolled studies and were liable to some uncertainty; even in some rare randomized controlled trials, the conclusions were contradictory. Moreover, adhesive ileus is just one variant of mechanical ileus; some researchers have pointed out the MIS can paradoxically create some specific types of mechanical ileus, such as internal or external herniation of small intestine, or bowel twisting over the anastomotic site, and so on. Therefore, it remains unclear whether MIS colorectal resection can reduce the incidence of the mechanical ileus and improve the long-term bowel function, as compared with the TOS.

Considering the aforementioned reasons, we conducted the present study to investigate if the incidence, patterns and the treatment outcomes of post-operative mechanical ileus changed in the era of MIS for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients whose primary colorectal cancers were resected in the fashion of curative and elective surgery.

Exclusion Criteria:

* patients who underwent palliative or emergency surgery to treat their primary colorectal cancer;
* patients encountered anastomotic leakage, intra-abdominal abscess or the other surgical complications requiring an additional abdominopelvic surgical or non-surgical procedures to treat the complications;
* simultaneously underwent some other abdominal or pelvic surgical procedures before or after the primary colorectal surgery, e.g., reverse Hartmann's procedure or closure of the temporary colostoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who diagnosed as colorectal cancer and underwent curative intent surgery
Sampling Method: Non-Probability Sample
Enrollment: 1544 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
Onset time | Follow up period about five years with a median of 38.5 months.
  Patients with mechanical ileus were stratified as acute, early, intermediate, and late onset, according to whether the mechanical ileus occurred within 3 months, 3-12 months, 1-2 years, or more than 2 years after the primary surgery for colorectal cancer, respectively.

SECONDARY OUTCOMES:
The pattern of adhesion | Follow up period about five years with a median of 38.5 months.
  The pattern of adhesion may be recorded as follows: bands (>1 cm long and <1 cm diameter); simple adhesions (<1 cm long and >1 cm diameter) or matted adhesion (dense, multiple, and tangled)
The surgery of adhesive ileus | Follow up period about five years with a median of 38.5 months.
  The surgery for treating ileus may be recorded as follows: 1) band section; 2) lysis of simple adhesion; 3) lysis of matted adhesion; 4) extensive adhesiolysis, sutured or not serosal defect or sutured accidental enterotomies; or 5) even the segmental bowel resection in addition to whatever the previously mentioned procedures.
Blood loss | About 3-4 hours
  The intraoperative blood loss was recorded in mL.
Operation time | About 3-4 hours
  The operation time was recorded in minutes.
Surgical complication | Within 30 days
  The Clavien-Dindo classification system was used to score the severity of surgical complications. The Clavien-Dindo Classification consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The higher the grade, the severer the complication.
Hospitalization | About 7-10 days
  The length of hospital stay was calculated from the date of surgery for mechanical ileus to the day of discharge from the hospital.
Re-admission | Within 30 days
  The patient needs to be readmitted to hospital due to index surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung LIANG, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided